CLINICAL TRIAL: NCT06924320
Title: A Phase 1 Randomized, Double-Blind, Placebo Controlled. Single and Multiple Ascending Dose Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of MET233 Co-administered With MET097 in Adult Participants With Obesity or Overweight Including Participants With Type 2 Diabetes Mellitus
Brief Title: A Study of MET233 in Combination With MET097 in Individuals With Obesity or Overweight With or Without Diabetes
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Metsera, a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MET233/097-24-101
Record Dates: First submitted 2025-04-03; First posted 2025-04-11 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Obesity and Obesity-related Medical Conditions
Keywords: GLP-1; Metsera
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- SAD: MET233 co-administered with MET097 (Experimental): Participants in the single ascending dose cohorts will receive subcutaneous MET233 co-administered with MET097 at a single point in time.
  Interventions: Drug: MET233 and MET097
- SAD: Placebo (Placebo Comparator): Participants in the single ascending dose cohorts will receive subcutaneous Placebo at a single point in time.
  Interventions: Drug: Placebo
- MAD: MET233 co-administered with MET097 (Experimental): Participants in the multiple ascending dose cohorts will receive subcutaneous MET233 co-administered with MET097 weekly.
  Interventions: Drug: MET233 and MET097
- MAD: Placebo (Placebo Comparator): Participants in the multiple ascending dose cohorts will receive subcutaneous Placebo weekly.
  Interventions: Drug: Placebo
- MAD: MET233 co-administered with Placebo (Experimental): Participants will receive subcutaneous MET233 co-administered with Placebo weekly.
  Interventions: Drug: MET233

INTERVENTIONS:
Drug: MET233 and MET097 — For subcutaneous administration
  Arms: MAD: MET233 co-administered with MET097; SAD: MET233 co-administered with MET097
Drug: Placebo — Sterile 0.9% (w/v) saline for subcutaneous administration.
  Arms: MAD: Placebo; SAD: Placebo
Drug: MET233 — For subcutaneous administration
  Arms: MAD: MET233 co-administered with Placebo

SUMMARY:
This study is designed to test how well the combination of MET233 with MET097 works to treat individuals with obesity or overweight with or without diabetes.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, double-blind, double-dummy study to investigate the safety, tolerability, PK, and PD of subcutaneous (SC) doses of MET233 co-administered with MET097 in adult participants with a BMI of 27 to 38 kg/m2, including some participants with T2DM. For Part A, after the up to 4-week screening period, the study includes 1 dose and a 12-week safety follow-up after administration. For Part B and Part C, after the up to 4-week screening period, the study includes 12 once-weekly doses and an approximately 11-week safety follow-up after the last administration. Parts A and B will include only participants with overweight or obesity without type 2 diabetes. Part C will include participants with overweight or obesity who also have type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥27 kg/m2 and ≤38.0 kg/m2 (inclusive) at screening
* For participants in Part A and B, no history of clinically significant diseases or clinically significant findings from the physical examination. For participants in Part C, no clinically significant diseases except T2DM, well controlled hypertension, and/or dyslipidemia.
* For participants in Part C, diagnosed with T2DM for at least 3 months before screening.
* For participants in Part C, T2DM includes glycated hemoglobin (HbA1c) value ≤10.5% at Screening and treated with stable therapy for at least 30 days prior to Screening/Visit 1.

Exclusion Criteria:

* Female who is lactating or who is pregnant according to the pregnancy test at Screening or on Day 1.
* Seated blood pressure higher than 160/100 mmHg at the Screening visit or prior to the first study drug administration.
* Elevated resting pulse greater than 100 beats per minute at Screening visit or prior to the first study drug administration.
* Estimated glomerular filtration rate (eGFR) <80 mL/min at the Screening visit.
* Diagnosis of Type 1 diabetes.
* For Part A and Part B: Diagnosis of T2DM or glycated hemoglobin (HbA1c) > 6.4% or fasting plasma glucose >126 mg/dL at the Screening visit or history of taking any medications to lower glucose.
* For Part A and Part B: Participant reported weight-related comorbidity, including sleep apnea and cardiovascular disease.
* History of bariatric or weight loss surgeries.
* Personal or family history of medullary thyroid carcinoma or multiple endocrine neoplasia syndrome.
* Lifetime history of acute or chronic pancreatitis or pancreatic cancer.
* Participation in a weight loss program with or without pharmacotherapy during the 3 months prior to study administration or plans to do so.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2027-01-25 (Estimated); Study Completion 2027-03-15 (Estimated)

PRIMARY OUTCOMES:
Part A: Occurrence of treatment-emergent adverse events (TEAEs) | Baseline (Week 0) to Day 85 (Week 12)
Part B: Occurrence of treatment-emergent adverse events (TEAEs) | Baseline (Week 0) to Day 155 (Week 22)
Part C: Occurrence of treatment-emergent adverse events (TEAEs) | Baseline (Week 0) to Day 155 (Week 22)

SECONDARY OUTCOMES:
Part A: Maximum observed concentration (Cmax) | Baseline (Week 0 ) through Day 85 (Week 12)
Part B: Maximum observed concentration (Cmax) | Baseline (Week 0 ) through Day 155 (Week 22)
Part C: Maximum observed concentration (Cmax) | Baseline (Week 0 ) through Day 155 (Week 22)
Part A: Area under the concentration versus time curve (AUC) | Baseline (Week 0 ) through Day 85 (Week 12)
Part B: Area under the concentration versus time curve (AUC) | Baseline (Week 0 ) through Day 155 (Week 22)
Part C: Area under the concentration versus time curve (AUC) | Baseline (Week 0 ) through Day 155 (Week 22)
Part A: Time to maximum observed concentration (Tmax) | Baseline (Week 0 ) through Day 85 (Week 12)
Part B: Time to maximum observed concentration (Tmax) | Baseline (Week 0 ) through Day 155 (Week 22)
Part C: Time to maximum observed concentration (Tmax) | Baseline (Week 0 ) through Day 155 (Week 22)
Part A: Minimum observed concentration (Cmin) | Baseline (Week 0 ) through Day 85 (Week 12)
Part B: Minimum observed concentration (Cmin) | Baseline (Week 0 ) through Day 155 (Week 22)
Part C: Minimum observed concentration (Cmin) | Baseline (Week 0 ) through Day 155 (Week 22)
Part A: Percent change from baseline in body weight | Weekly post-baseline up to Day 85 (Week 12)
Part B: Percent change from baseline in body weight | Weekly post-baseline up to Day 155 (Week 22)
Part C: Percent change from baseline in body weight | Weekly post-baseline up to Day 155 (Week 22)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Research Site MET233/097 24-101-001, Cypress, California, United States